CLINICAL TRIAL: NCT00417131
Title: Imaging of Islet Transplantation With PET and MRT
Status: Completed | Type: Observational
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Gunnar Tufveson, MD, Professor, Uppsala University Hospital
Other Study IDs: Studieprotokoll 2006-05-12
Record Dates: First submitted 2006-12-28; First posted 2006-12-29 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2008-07

CONDITIONS: Islet Transplantation; Diabetes Type 1
Keywords: Islet transplantation,; coagulation,; graft destruction,; islet imaging
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Islets of Langerhans intended for clinical transplantation are labelled with a radioactive tracer. The tracer is retained in viable cells of the transplant. At infusion (transplantation) of the islets into the portal vein the tracer can be followed for two hours with positron emission tomography (PET). Imaging and calculations can give estimates of the proportion of surveying islets and the rate of early destruction. Also the distribution of the islets into the liver can be viewed.

DETAILED DESCRIPTION:
Background:

It is suspected that the current need for repeated islets transplantation to treat diabetes type I is dependent on an early destruction of the islets when infused into the portal vein.

Aim:

To trace the fate of the islet at and after infusion into the portal vein.

Method:

Islets are labelled in vitro with a radioactive tracer that can be measured with positron emission tomography. 10-20 percent of the graft is labelled. Just prior to start of infusion labelled islets are mixed with unlabelled islets (80-90 percent of the graft). The tracer used is FDG and stands for 2-[18F]-2-deoxy-D-glucose. At infusion the patient is placed in the combined computer tomography and PET camera to follow the infusion. The imaging is almost continuous for 2 h at and after infusion.

Expected results:

Calculations of proportion of surviving islets and rate of destruction. Localisation and distribution of islets in the liver of the recipient.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for clinical islet transplantation.
* Patient on waiting list for islet transplantation within the Nordic Network for Clinical Islet Transplantation
* Written Informed Concent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients referred to islet transplantation in the Nordic countries (Scandinavia)
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2006-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Tufveson, Professor, Principal Investigator — Dept of Transplantation, Uppsala University Hospital
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Dept. of Transplantation surgery, Stockholm
  - Uppsala University Hospital, Dept of Transplantation Surgery, Uppsala

REFERENCES:
- [Derived] Eriksson O, Eich T, Sundin A, Tibell A, Tufveson G, Andersson H, Felldin M, Foss A, Kyllonen L, Langstrom B, Nilsson B, Korsgren O, Lundgren T. Positron emission tomography in clinical islet transplantation. Am J Transplant. 2009 Dec;9(12):2816-24. doi: 10.1111/j.1600-6143.2009.02844.x. Epub 2009 Oct 21. PMID 19845588